CLINICAL TRIAL: NCT05610917
Title: Construction and Evaluation of Risk Early Warning Mechanism of Physical Cognitive Decline Syndrome and Community-based Rehabilitation Management Program for Patients With Remitted Geriatric Depression
Brief Title: Community-based Rehabilitation Management for Patients With Remitted Geriatric Depression
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Duan Li (Other)
Responsible Party: Sponsor-Investigator, Duan Li, Doctor Duan, Chengde Medical University
Organization: Chengde Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChengdeMU
Record Dates: First submitted 2022-10-27; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Geriatric Depression
Keywords: Remitted geriatric depression; Physio-cognitive decline syndrome; risk early warning mechanism; community-based rehabilitation management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case group, (Experimental): Patients in case group will be treated with CBRM program
  Interventions: Combination Product: CBRM (community-based rehabilitation management)
- control group (Other): the control group patients will be treated routinely as usual.
  Interventions: Combination Product: TAR(treatment as routine)

INTERVENTIONS:
Combination Product: CBRM (community-based rehabilitation management) — The case group patients will undergo drug treatment (Selective Serotonin Reuptake Inhibitors), health education, cognitive-motor dual task training, cognitive-training.
  Arms: case group,
Combination Product: TAR(treatment as routine) — Patients in control group will be treated rountinely which includes drug treatment (SSRIs) and traditional health education.
  Arms: control group

SUMMARY:
This study intends to take patients with RGD as objects. Further construct a community-based rehabilitation management (CBRM) program with drug treatment, rehabilitation measures of education, psychology and exercise as its core content on the basis of evidence-based practice approach. Based on the cost-utility analysis of health economics, the health and economic benefits of the CBRM program will be evaluated, and a theoretical reference will be provided for community health institutions to carry out whole-course rehabilitation management practice and health policy formulation.

DETAILED DESCRIPTION:
Based on the background of population aging, the prevalence of Late life depression tends to increase, and the recurrence rate after antidepressants treatment is still as high as 35%-57%, and the disease course tends to be chronic. Therefore, the formulation and implementation of prevention and control programs have become a significant part of the government's work plan. Physical frailty symptoms such as loss of daily activities and weakness are common in patients with remitted geriatric depression (RGD), and cognitive impairment is also considered to be an independent persistent symptom of RGD patients, which are related to the fluctuation and recurrence of depressive symptoms in elderly patients. Physical cognitive decline syndrome (PCDS) can comprehensively assess the physical frailty symptoms and the degree of cognitive impairment of the elderly, and effectively predict the course of the disease and the trend of healthy development. However, studies applied to the field of emotional disorder have not been retrieved. Therefore, this study intends to take patients with RGD as objects to investigate the prevalence of PCDS, build a risk prediction model and reveal it is warning mechanisms. That is, after determinning the basis of risk factors affecting the occurence of PCDS in RGD patients, we will carry out the formulation, implementation and evaluation of the follow-up CBRM program.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years old or above at the time of enrollment;
* meet the diagnostic criteria for MDD without psychotic features according to DSM-5, and depressive symptoms have been improved and remained stable for at least 2 months after treatment with SSRIs;
* the total score of HAMD-17 is less than 7 at the time of enrollment;
* meet the diagnostic criteria for physio-cognitive decline: 1) the total score of ADL and IADL was less than 26; 2)cognitve decline: first, subjects with severe impairment of cognitive function will be excluded (years of education ≥ 6, MMSE scores <24；years of education <6 years, MMSE total score <14). After completing a neuropsychological task, cogintive declined will be confirmed when any aspects of cognitve function is 1.5 standard deviations lower than that of normal elderly; 3) the grip strength is weakened, and the domaint hand grip strength is < 28kg for males or <18kg for females; 4)slow step speed, that is, in a space of length >10 meters, the subjects walks 6 meters from the starting point at a normal and uniform pace, and the pace is <1m/s.
* comprehension, reading and writing skills to complete the measurements or complete them with assistance of the researchers with obstacles;
* voluntary participation and signed informed consent.

Exclusion Criteria:

* meet the diagnostic of schizophrenia, bipolar disorder, dementia;
* comorbidity of physical diseases, such ascardiovascular and cerebrovascular diseases, rheumatoid arthritis, stroke and malignant tumors;
* history of alcohol or drug dependence;
* severe deformity of spine and limbs;
* complete or partial dependence on caregivers for daily life, such as long-term bedridden, wheelchair assisted;
* have received physical therapy or psychological treatment in the past three months;
* currently participating in other clinical research.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
depressive symptoms | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  The Hamilton Depressive Scale (HAMD-17) which consists of 17 items will be employed to screen for depressive symptoms and evaluate the mental status and severity of depressive symptoms. Scores were calculated by totaling the responses, which can be divided into four types (Health): normal/not depressed (0-7 points), mild/subthreshold (8-13), moderate/mild (14-18), severe/moderate (19-22), and severe/very severe (>23).
cognitive and intellectual function | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  Mini-mental State Examination (MMSE), as a simple screening tool for cognitive and intellectual function decline in the elderly with a total score of 30. The results of this test is closely related to the level of education, and the normal cutoff is defined as, illiterates >17 points, primary schools >20 points, and middle schools and above >24 points.
changes of the handgrip strength | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  The grip strength of a man's dominant hand < 28kg or a woman < 18kg is considered to have weak grip strength. The grip strength increased compared with the baseline period, that is, the subjects' physiological function tended to recover; Instead, physiological function tends to decline.
changes of the gait speed | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  The time it takes for the subject to walk 6 meters at normal pace from the starting point without slowing down, with a threshold for gait deceleration set to < 1m/s. The gait speed increased compared with the baseline period, that is, the subjects' physiological function tended to recover; Instead, physiological function tends to decline.

SECONDARY OUTCOMES:
quality of life of the elderly | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  The WHO Quality of Life Scale (WHOQOL-BREF Chinese version) includes four dimensions, such as physiological, psychological, social relations and environment, covering 26 items related to quality of life. This scale is widely used in patients with cancer, chronic diseases and the elderly. Each item is scored according to Likert 1-5. The higher the total score, the better the quality of life.
sleep quality | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  The Pittsburgh Sleep Quality Index (PSQI) will be used to measure the subjects' sleep treatment. The total score range is 0-21 points. It is generally believed that the total score of PSQI ≤7 indicates that the sleep quality is fair, while the total score of > 7 indicates poor sleep quality, and the higher the total score of PSQI scale, the worse the sleep quality of the subjects.
the balance ability of the elderly | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  The Short Physical Performance Battery test (SPPB) will be used to assess the balance ability of the elderly, including: (1) Sit-stand test for 5 times. The shorter the time, the better the balance ability. (2) Timing test of 2.44m short distance walking. The shorter the time, the better the balance ability. (3) Balance function test, the longer the time, the better the balance ability.
activity of daily living | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  Activity of Daily Living (ADL) whose total score is ranging from 14 to 56. Total score ≤26, basically normal; > 26 indicates different degree of functional decline; Score of 2 or more individual scores > 3 points, significant dysfunction.
the word memory function | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  Chinese Version Verbal Learning Test (CVVLT) will be used to evaluate the word memory function of the elderly. Researchers repeated 9 words at a rate of one word per second for four times in a fixed sequence. The elderly will be asked to recall the words 30 seconds later and again 10 minutes later. In this study, only the results of the delayed free memory test at the 10th minute will be included in the later statistics. The more vocabularies remembered, the better the cognitive function.
language functions | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  Boston Naming Test (BNT-30) will be used to evaluate language functions of the elderly. During the test, if the subject could make a spontaneous naming error within 20 seconds, the semantic cue will be used to prompt the subject; if the subject could not answer within 20 seconds, the subject will be given a recognition choice including three choices. The evaluation indexes include spontaneous correct naming number, prompt correct naming percentage and selection of correct naming percentage. The higher the score, the better the cognitive function.
verbal functions | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  Verbal Fluency Test (VFT) will be used to assess the verbal functions of the elderly. Subjects are required to say as many animal names as possible within one minute. The test involves multiple cognitive functions such as memory, language and execution, which is the most important tool for testing subjects' language fluency. The more words they can say, the better their cognitive function.
visuospatial structure ability and visual memory of the elderly | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  Rey-Osterrieth Complex Figure Test (ROCFT) will be used to asses the visuospatial structure ability and visual memory of the elderly. During the test, the elderly will be asked to copy complex images. Researchers record the copying time and remove the cards immediately after the copying completed. After 3 minutes and 30 minutes, the subjects will be asked to re-draw according to the recall, and the researchers record the duration of the instantaneous recall. Each drawing should take no more than 10 minutes. Reference standards will used to score the images of copying, instantaneous meeting and delayed recall respectively, with a total score of 36 points.
working memory portion of the executive function | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  Digital Backward (DB) will be used to evaluate the working memory portion of the executive function. The elderly will be asked to read a sequence of numbers at a rate of one number per second and asked to immediately repeat the sequence in reverse order. The number of numbers in the last sequence that the subject can recite correctly is the score of the DB test.
the executive ability and the visuospatial ability | This variable will be measured at 0 (baseline) and after 3, 6 months post-intervention.
  Clock Drawing Test (CDT) will be used to evaluate the executive ability and the visuospatial ability. Subjects will be asked to draw the face of a clock and write all the numbers. The hour and minute hands point to 11:10. The clock face is complete (0-2 points), the number is complete and sequence (0-4 points), and the pointer is complete and position (0-4 points). The higher the total score is, the better the cognitive function is.

CONTACTS AND LOCATIONS:
Overall Officials: Li Duan, Dr., Study Director — Chengde Medical University
Locations (1):
- Chengde Medical University, Chengde, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen LK, Arai H. Physio-cognitive decline as the accelerated aging phenotype. Arch Gerontol Geriatr. 2020 May-Jun;88:104051. doi: 10.1016/j.archger.2020.104051. Epub 2020 Apr 4. No abstract available. PMID 32278485
- [Result] Liu LK, Chou KH, Hsu CH, Peng LN, Lee WJ, Chen WT, Lin CP, Chung CP, Wang PN, Chen LK. Cerebellar-limbic neurocircuit is the novel biosignature of physio-cognitive decline syndrome. Aging (Albany NY). 2020 Nov 25;12(24):25319-25336. doi: 10.18632/aging.104135. Epub 2020 Nov 25. PMID 33234736
- [Result] Liang CK, Lee WJ, Hwang AC, Lin CS, Chou MY, Peng LN, Lin MH, Chen LK. Efficacy of Multidomain Intervention Against Physio-cognitive Decline Syndrome: A Cluster-randomized Trial. Arch Gerontol Geriatr. 2021 Jul-Aug;95:104392. doi: 10.1016/j.archger.2021.104392. Epub 2021 Mar 13. PMID 33765656
- [Result] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Result] Chen LK, Hwang AC, Lee WJ, Peng LN, Lin MH, Neil DL, Shih SF, Loh CH, Chiou ST; Taiwan Health Promotion Intervention Study for Elders research group. Efficacy of multidomain interventions to improve physical frailty, depression and cognition: data from cluster-randomized controlled trials. J Cachexia Sarcopenia Muscle. 2020 Jun;11(3):650-662. doi: 10.1002/jcsm.12534. Epub 2020 Mar 5. PMID 32134208
- [Result] Merchant RA, Chan YH, Hui RJY, Tsoi CT, Kwek SC, Tan WM, Lim JY, Sandrasageran S, Wong BLL, Chen MZ, Ng SE, Morley JE. Motoric cognitive risk syndrome, physio-cognitive decline syndrome, cognitive frailty and reversibility with dual-task exercise. Exp Gerontol. 2021 Jul 15;150:111362. doi: 10.1016/j.exger.2021.111362. Epub 2021 Apr 19. PMID 33887381